CLINICAL TRIAL: NCT01853722
Title: A Phase 2, Open-Label, Randomized, Parallel Group, Placebo-Controlled, Single-Center Study to Assess Anti-microbial Efficacy and Safety of DCN01 Compared to Unisol® Following Topical Periocular Administration in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deacon Biosciences, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-150-0002
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Ocular Infection
Keywords: DCN01; Ocular Surgical Preparation; Prophylaxis against infection; Pre-operative prep
MeSH Terms: conditions — Eye Infections | interventions — UHK solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCN01 (Experimental)
  Interventions: Drug: DCN01
- Unisol (Placebo Comparator)
  Interventions: Drug: Unisol

INTERVENTIONS:
Drug: DCN01 — Three serial applications per periocular region.
  Arms: DCN01
Drug: Unisol — Three serial applications per periocular region.
  Arms: Unisol

SUMMARY:
This proof-of-concept study evaluates the clinical efficacy and safety of DCN01 in prepping of the periocular region.

ELIGIBILITY:
Inclusion Criteria:

* Have given a written, informed consent
* Be willing and able to follow all instructions
* A negative urine pregnancy test if female of childbearing potential

Exclusion Criteria:

* Known sensitivities to study medication or its components
* Any signs of an active infection
* Use of disallowed products during the period indicated prior to the enrollment or during the study
* Be currently pregnant, nursing, or planning a pregnancy; or be a woman that has a positive pregnancy test
* Have a condition or a situation which, in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in periocular region bacterial load | Baseline to 10 min post dose

SECONDARY OUTCOMES:
Proportion of periocular regions with a reduction from baseline in bacterial load. | Baseline to 10 min post dose

OTHER OUTCOMES:
Adverse Events (reported, elicited, observed) | Post dose and up to 2 weeks after (Day 1-14)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States